CLINICAL TRIAL: NCT04418492
Title: An Intervention Program Targeting Daily Adaptive Skills Through Executive Function Training for Adults With Autism Spectrum Disorder: A Pilot Study
Brief Title: An Intervention Targeting Daily Adaptive Skills Through Executive Function Training for Adults With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1904/537-302
Record Dates: First submitted 2020-05-21; First posted 2020-06-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Autism Spectrum Disorder; High-functioning Autism; Autism
Keywords: Autism Spectrum Disorder; High-functioning Autism; Autism; Executive Function; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAFE intervention (Experimental): The single group received the SAFE intervention for 10 weeks.
  Interventions: Behavioral: Skills for Adaptive Functioning through Executive training (SAFE; tentative title)

INTERVENTIONS:
Behavioral: Skills for Adaptive Functioning through Executive training (SAFE; tentative title) — An intervention program to improve adaptive skills and executive functions in young adults with high-functioning autism spectrum disorder was administered weekly for 10 weeks to the participants. The participants also completed pre-, mid- and post-intervention assessments.

SUMMARY:
The current study is a single group pilot study of a novel intervention program which targets improvements in executive functions and adaptive skills in transition age young adults with high-functioning autism spectrum disorder. The main aim of the study is to test the effectiveness of the intervention using a pretest-posttest comparison. It is hypothesised that there will be an increase in executive functions and adaptive skills after the intervention.

DETAILED DESCRIPTION:
The participants engaged in a 10-week group-based intervention program which aims to improve daily adaptive skills based on executive functions and help the transition into adulthood in young adults with ASD. Before and after the intervention, the participants and their parents completed questionnaires that measure executive functions and adaptive skills, and the participants additionally completed an assessment of social adaptive skills. The differences between pre- and post-intervention scores of the outcome measures were analyzed using Wilcoxon signed-rank tests to evaluate the effect of the program.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of ASD as measured by the Autism Diagnostic Observation Schedule and the Autism Diagnostic Interview-Revised
* Full-scale IQ of 70 or above as measured by the Weschler Adult Intelligence Scale

Exclusion Criteria:

* Full-scale IQ less than 70
* Uncooperative and lacking motivation to participate in the programme
* Reporting clinically significant behavioural problems, emotion regulation problems, psychotic symptoms, risk of self-harm or harm to others which can affect the participation to the programme, which is screened by the screening assessments and interviews.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
The change in the Korean version of Barkley Deficits in Executive Functioning Scale (K-BDEFS) | 1 week before the intervention, between 5th and 6th session of the intervention and 1-3 week after the intervention.
  The Korean version of Barkley Deficits in Executive Functioning Scale measures executive functions of adults in everyday life. The score range is 89-356. Higher score indicates worse executive functioning.
The change in the Korean version of Vineland Adaptive Behavior Scale-II (K-Vineland-II) | 1 week before the intervention and 1-3 week after the intervention.
  The Korean version of Vineland Adaptive Behavior Scale-II measures adaptive behavior. The scores are converted into a standard score with a mean of 100 and a standard deviation of 15. Higher score indicates better adaptive functioning.
The change in the Community Integration Skills Assessment-2 (CISA-2) | 1 week before the intervention and 1-3 week after the intervention.
  The Community Integration Skills Assessment-2 measures adaptive skills necessary for people with developmental disorders to integrate into the community. The scores are converted into a standard score with a mean of 100 and a standard deviation of 15. Higher score indicates better community integration skills.
The change in the Cognitive Flexibility Inventory (CFI) | 1 week before the intervention and 1-3 week after the intervention.
  The Cognitive Flexibility Inventory assesses cognitive flexibility. The score range is 19-113. Higher score indicates better cognitive flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jeong Yoo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No